CLINICAL TRIAL: NCT04896086
Title: VRC 325 (000410): A Phase I Open-Label Clinical Trial to Evaluate the Dose, Safety, Tolerability and Immunogenicity of Mosaic Quadrivalent Influenza Vaccine With and Without Adjuplex Compared With a Licensed Inactivated Seasonal QIV, In Healthy Adults
Brief Title: First-in-Human Clinical Trial of a Mosaic Quadrivalent Influenza Vaccine Compared With a Licensed Inactivated Seasonal QIV in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10000410; 000410-I
Record Dates: First submitted 2021-05-20; First posted 2021-05-21 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Influenza; Seasonal Influenza
Keywords: Seasonal Influenza; Flu Virus; Respiratory Illness; Viral Infection; Experimental Vaccine; Nanoparticle Vaccine; Adjuvant
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) (Experimental): FluMos-v1 (20 mcg) administered intramuscularly (IM) by needle/syringe
  Interventions: Drug: VRC-FLUMOS0111-00-VP (FluMos-v1)
- Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) (Experimental): FluMos-v1 (60 mcg) administered intramuscularly (IM) by needle/syringe
  Interventions: Drug: VRC-FLUMOS0111-00-VP (FluMos-v1)
- Part A, Group 3 (3A-3B): Flucelvax (60 mcg) (Active Comparator): Licensed QIV Flucelvax (60 mcg) administered intramuscularly (IM) by needle/syringe
  Interventions: Biological: Flucelvax
- Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) (Experimental): FluMos-v1 (100 mcg) administered intramuscularly (IM) by needle/syringe
  Interventions: Drug: VRC-FLUMOS0111-00-VP (FluMos-v1)
- Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v) (Experimental): FluMos-v1 (100 mcg) plus Adjuplex (20% v/v) administered intramuscularly (IM) by needle/syringe
  Interventions: Drug: VRC-GENADJ0110-AP-NV (Adjuplex); Drug: VRC-FLUMOS0111-00-VP (FluMos-v1)

INTERVENTIONS:
Drug: VRC-GENADJ0110-AP-NV (Adjuplex) — Adjuplex is a sterile, pyrogen-free adjuvant solution produced by the VRC Pilot Plant. Adjuplex comprises highly purified de-oiled soy lecithin and benzene-free carbomer homopolymer formulated in phosphate buffered saline. Adjuplex adjuvant was mixed with FluMos-v1 at 20% by volume in the pharmacy during product preparation for the vaccinations of Groups 5A-5B.
  Other Names: Adjuplex
  Arms: Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Biological: Flucelvax — Flucelvax is an inactivated influenza vaccine licensed for the 2020-2021 season.
  Arms: Part A, Group 3 (3A-3B): Flucelvax (60 mcg)
Drug: VRC-FLUMOS0111-00-VP (FluMos-v1) — FluMos-v1 investigational vaccine is composed of engineered pentameric promoters based on C. albicans lumazine synthase assembled with 20 trimeric promoters displaying HA ectodomains. It contains hemagglutinin (HA) proteins from the following 4 influenza strains: A/Idaho/07/2018, A/Perth/1008/2019, B/Colorado/06/2017 and B/Phuket/3073/2013.
  Other Names: FluMos-v1
  Arms: Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg); Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg); Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg); Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)

SUMMARY:
Background:

Influenza (flu) is a contagious respiratory illness. It is caused by influenza viruses that infect the nose, throat, and sometimes the lungs. Vaccines are given to teach the body to prevent or fight infection. Researchers want to study a new vaccine to prevent the seasonal flu.

Objective:

To see if the FluMos-v1 vaccine is safe and how the body responds to it.

Eligibility:

Healthy adults ages 18-50 years inclusive were enrolled.

Design:

Participants were screened through a separate protocol.

Participants were tested for COVID-19. They may have had a pregnancy test.

Participants received the investigational FluMos-v1 vaccine or the licensed inactivated seasonal quadrivalent influenza vaccine Flucelvax injected in the upper arm.

Participants completed a diary card for 7 days. They recorded any symptoms they had. They were given a thermometer to check their temperature. They were also given a ruler to measure any skin changes at the injection site.

Participants had about 10 study visits. They were asked how they were feeling and if they had taken any medications. They had blood drawn.

Some participants had an optional apheresis. Blood was removed through a needle in a vein in one arm. A machine separated the white blood cells. The rest of the blood was returned through a needle in a vein in the other arm.

Participation lasted for 40 weeks.

DETAILED DESCRIPTION:
Design:

This was a Phase I, open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of the mosaic quadrivalent influenza vaccine VRC-FLUMOS0111-00-VP (FluMos-v1). The hypotheses were that the FluMos-v1 vaccine is safe and tolerable and would elicit an immune response. The primary objective was to evaluate the safety and tolerability of the investigational vaccine alone or with adjuvant in healthy adults. Secondary objectives were related to immunogenicity of the investigational vaccine and dosing regimen compared with the licensed inactivated seasonal Flucelvax (Registered Trademark) quadrivalent influenza vaccine (QIV) in healthy adults.

Study Products:

The investigational nanoparticle vaccine VRC-FLUMOS0111-00-VP (FluMos-v1) was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID). FluMos-v1 is composed of engineered pentameric promoters based on C. albicans lumazine synthase assembled with 20 trimeric promoters displaying HA ectodomains. It contains hemagglutinin (HA) proteins from the following 4 influenza strains: A/Idaho/07/2018, A/Perth/1008/2019, B/Colorado/06/2017 and B/Phuket/3073/2013. FluMos-v1 was supplied in a single-use vial at a concentration of 180 mcg/mL.

In Part A, FluMos-v1 was compared to licensed 2020-2021 QIV Flucelvax (Registered Trademark) that was developed by Seqirus, Inc. and formulated with the following 4 influenza strains: A/Hawaii/70/2019 (H1N1) pdm09-like virus, A/Hong Kong/45/2019 (H3N2)-like virus, B/Washington/02/2019-like virus, and B/Phuket/3073/2013-like virus.

In Part B, a higher dose of FluMos-v1 was tested that more closely matches the amount of each HA antigen in Flucelvax. The adjuvant Adjuplex (Registered Trademark) was added to FluMos-v1 to evaluate the potential for increased immunogenicity.

Adjuplex is a sterile, pyrogen-free adjuvant solution produced by the VRC Pilot Plant. Adjuplex comprises highly purified de-oiled soy lecithin and benzene-free carbomer homopolymer formulated in phosphate buffered saline at a pH of 6.5 plus or minus 0.3. Adjuplex was provided as a sterile, pyrogen-free, homogeneous solution filled to 0.7 mL in 3-mL glass vials. Adjuplex was mixed with study products in the pharmacy during preparation prior to vaccination at a 20% dose by volume.

FluMos-v1, FluMos-V1 plus Adjuplex, and Flucelvax were administered intramuscularly (IM) in the deltoid muscle via needle and syringe.

Participants:

A total of 63 participants enrolled as follows:

Part A

Part A, Group 1 (20 mcg FluMos-v1): 5 participants

Group 1A (N=1): Did not receive 2020-2021 season's licensed influenza vaccine at any time prior to enrollment

Group 1B (N=4): Receipt of the 2020-2021 season's licensed influenza vaccine more than 4 months prior to enrollment

Part A, Group 2 (60 mcg FluMos-v1): 15 participants

Group 2A (N=4): Did not receive 2020-2021 season's licensed influenza vaccine at any time prior to enrollment

Group 2B (N=11): Receipt of the 2020-2021 season's licensed influenza vaccine more than 4 months prior to enrollment

Part A, Group 3 (60 mcg Flucelvax®): 15 participants

Group 3A (N=3): Did not receive 2020-2021 season's licensed influenza vaccine at any time prior to enrollment

Group 3B (N=12): Receipt of the 2020-2021 season's licensed influenza vaccine more than 4 months prior to enrollment

Part B

Part B, Group 4 (100 mcg FluMos-v1): 15 participants

Group 4A (N=1): Did not receive 2021-2022 or 2022-2023 season's licensed influenza vaccine at any time prior to enrollment

Group 4B (N=14): Receipt of the 2021-2022 or 2022-2023 season's licensed influenza vaccine more than 4 months prior to enrollment

Part B, Group 5 (100 mcg FluMos-v1 + Adjuplex (20% v/v)): 13 participants

Group 5A (N=2): Did not receive 2021-2022 or 2022-2023 season's licensed influenza vaccine at any time prior to enrollment

Group 5B (N=11): Receipt of the 2021-2022 or 2022-2023 season's licensed influenza vaccine more than 4 months prior to enrollment

Study Plan:

In Part A, the study evaluated the safety, tolerability, and immunogenicity of a single dose of FluMos-v1 vaccine alone in a dose-escalation design.

In Part B, the study evaluated the safety, tolerability, and immunogenicity of a single dose of FluMos-v1 vaccine with or without Adjuplex.

Group 6 and Part C were optional, and a decision was made not to enroll the optional Groups 6-8 in the study.

The protocol required 1 vaccination visit, about 8 follow-up visits, and a telephone contact on the day after vaccination. Solicited reactogenicity were evaluated using a 7-day diary card. Assessment of vaccine safety included clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

Study Duration:

Participants were evaluated for 40 weeks following vaccine administration including through an influenza season.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participant must have met all of the following criteria:

1. Healthy adults between the ages of 18-50 years inclusive
2. Based on history and physical examination, in good general health and without history of any of the conditions listed in the exclusion criteria
3. Part A: Received at least one licensed influenza vaccine from 2016 through the 2019-2020 influenza season
4. Part B: Received at least one licensed influenza vaccine from 2017 through the 2022-2023 influenza season
5. Able and willing to complete the informed consent process
6. Available for clinic visits for 40 weeks after enrollment and through an influenza season
7. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
8. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) <=35 within the 56 days before enrollment

   Laboratory Criteria within 56 days before enrollment
9. White blood cells (WBC) and differential within institutional normal range or accompanied by the site Principal Investigator (PI) or designee approval
10. Total lymphocyte count >=800 cells/microliter
11. Platelets = 125,000 - 500,000 cells/microliter
12. Hemoglobin within institutional normal range or accompanied by the PI or designee approval
13. Alanine aminotransferase (ALT) <=1.25 x institutional upper limit of normal (ULN)
14. Aspartate aminotransferase (AST) <=1.25 x institutional ULN
15. Alkaline phosphatase (ALP) <1.1 x institutional ULN
16. Total bilirubin within institutional normal range or accompanied by the PI or designee approval.
17. Serum creatinine <=1.1 x institutional ULN
18. Negative for HIV infection by an FDA-approved method of detection

    Criteria applicable to women of childbearing potential:
19. Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on the day of enrollment
20. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through the end of the study

EXCLUSION CRITERIA:

Participant was excluded if one or more of the following conditions applied:

1. Breast-feeding or planning to become pregnant during the study

   Participant received any of the following substances:
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
3. Blood products within 16 weeks prior to enrollment
4. Live attenuated vaccines within 4 weeks prior to enrollment
5. Inactivated vaccines within 2 weeks prior to enrollment
6. Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
7. Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule
8. Current anti-TB prophylaxis or therapy
9. Previous investigational H1, H2, or H10 influenza vaccines, including Part A participants
10. Part A:

    1. Groups 1A, 2A, and 3A only: Receipt of the 2020-2021 season's licensed influenza vaccine at any time prior to enrollment
    2. Groups 1B, 2B, and 3B only: Receipt of the 2020-2021 season's licensed influenza vaccine within 4 months prior to enrollment.
11. Part B and C:

    1. Groups 4A and 5A only: Receipt of the 2021-2022 or 2022-2023 season's licensed influenza vaccine at any time prior to enrollment
    2. Groups 4B and 5B only: Receipt of the 2021-2022 or 2022-2023 season's licensed influenza vaccine within 4 months prior to enrollment.

    Participant had a history of any of the following clinically significant conditions:
12. Serious reactions to vaccines that preclude receipt of the study vaccination as determined by the investigator
13. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
14. Asthma that is not well controlled
15. Diabetes mellitus (type I or II), with the exception of gestational diabetes
16. Thyroid disease that is not well controlled
17. Idiopathic urticaria within the past year
18. Autoimmune disease or immunodeficiency
19. Hypertension that is not well controlled
20. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
21. Malignancy that is active or history of malignancy that is likely to recur during the period of the study
22. Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
23. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
24. Guillain-Barre Syndrome
25. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesia Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not shared because it has limited value in a small phase 1 trial of healthy volunteers. We instead report non-IPD (aggregate) data as required in ClinicalTrials.gov.

REFERENCES:
- [Background] Lambert LC, Fauci AS. Influenza vaccines for the future. N Engl J Med. 2010 Nov 18;363(21):2036-44. doi: 10.1056/NEJMra1002842. No abstract available. PMID 21083388
- [Background] Kanekiyo M, Joyce MG, Gillespie RA, Gallagher JR, Andrews SF, Yassine HM, Wheatley AK, Fisher BE, Ambrozak DR, Creanga A, Leung K, Yang ES, Boyoglu-Barnum S, Georgiev IS, Tsybovsky Y, Prabhakaran MS, Andersen H, Kong WP, Baxa U, Zephir KL, Ledgerwood JE, Koup RA, Kwong PD, Harris AK, McDermott AB, Mascola JR, Graham BS. Mosaic nanoparticle display of diverse influenza virus hemagglutinins elicits broad B cell responses. Nat Immunol. 2019 Mar;20(3):362-372. doi: 10.1038/s41590-018-0305-x. Epub 2019 Feb 11. PMID 30742080
- [Background] Boyoglu-Barnum S, Ellis D, Gillespie RA, Hutchinson GB, Park YJ, Moin SM, Acton OJ, Ravichandran R, Murphy M, Pettie D, Matheson N, Carter L, Creanga A, Watson MJ, Kephart S, Ataca S, Vaile JR, Ueda G, Crank MC, Stewart L, Lee KK, Guttman M, Baker D, Mascola JR, Veesler D, Graham BS, King NP, Kanekiyo M. Quadrivalent influenza nanoparticle vaccines induce broad protection. Nature. 2021 Apr;592(7855):623-628. doi: 10.1038/s41586-021-03365-x. Epub 2021 Mar 24. PMID 33762730
- [Background] Yang RS, Traver M, Barefoot N, Stephens T, Alabanza C, Manzella-Lapeira J, Zou G, Wolff J, Li Y, Resto M, Shadrick W, Yang Y, Ivleva VB, Tsybovsky Y, Carlton K, Brzostowski J, Gall JG, Lei QP. Mosaic quadrivalent influenza vaccine single nanoparticle characterization. Sci Rep. 2024 Feb 24;14(1):4534. doi: 10.1038/s41598-024-54876-2. PMID 38402303
- [Derived] Alabanza C, Gavrilov V, Scott T, Yang RS, Gowetski DB, Gall JG, Paula Lei Q. Quantitation of strain-specific hemagglutinin trimers in mosaic quadrivalent influenza nanoparticle vaccine by ELISA. Vaccine. 2023 Aug 7;41(35):5201-5210. doi: 10.1016/j.vaccine.2023.07.009. Epub 2023 Jul 12. PMID 37451877
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000410-I.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland.
Groups:
- Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v): FluMos-v1 (100 mcg) plus Adjuplex (20% v/v) administered intramuscularly (IM) by needle/syringe
  VRC-GENADJ0110-AP-NV: Adjuplex is a sterile, pyrogen-free adjuvant solution produced by the VRC Pilot Plant. Adjuplex comprises highly purified de-oiled soy lecithin and benzene-free carbomer homopolymer formulated in phosphate buffered saline. Adjuplex adjuvant was mixed with FluMos-v1 at 20% by volume in the pharmacy during product preparation for the vaccinations of Groups 5A-5B.
  VRC-FLUMOS0111-00-VP (FluMos-v1): FluMos-v1 investigational vaccine is composed of engineered pentameric promoters based on C. albicans lumazine synthase assembled with 20 trimeric promoters displaying HA ectodomains. It contains hemagglutinin (HA) proteins from the following 4 influenza strains: A/Idaho/07/2018, A/Perth/1008/2019, B/Colorado/06/2017 and B/Phuket/3073/2013.
Period: Overall Study
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Started | 5 | 15 | 15 | 15 | 13
Completed Product Administration | 5 | 15 | 15 | 13 | 13
Completed | 5 | 12 | 14 | 13 | 13
Not Completed | 0 | 3 | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Difficulties were experienced with vein access for blood sample collection | 0 | 0 | 0 | 1 | 0
Not completed — Participant had a syncopal event during a blood draw | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants. Age represents age at enrollment day. Height and weight (used for BMI) were from the enrollment evaluation per the eligibility criterion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v) | Total
Number analyzed (Participants) | 5 | 15 | 15 | 15 | 13 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] — Age represents age at enrollment day.
  years | 34.0 (11.1) | 27.3 (8.0) | 31.3 (7.8) | 28.7 (7.8) | 29.0 (7.3) | 29.5 (8.0)
Age, Customized [Count of Participants; unit: Participants] — Age represents age at enrollment day.
  Participants
    21-30 years | 2 | 10 | 8 | 10 | 9 | 39
    31-40 years | 2 | 4 | 5 | 4 | 3 | 18
    41-50 years | 1 | 1 | 2 | 1 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 8 | 9 | 5 | 32
  Male | 3 | 7 | 7 | 6 | 8 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 3 | 7
  Not Hispanic or Latino | 5 | 12 | 14 | 14 | 10 | 55
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 4 | 6 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 0 | 4
  White | 1 | 9 | 9 | 9 | 8 | 36
  More than one race | 1 | 2 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Height and weight (used for BMI) were from the enrollment evaluation per the eligibility criterion.
  kg/m^2 | 25.0 (2.1) | 23.6 (2.8) | 25.4 (3.8) | 23.0 (4.5) | 27.9 (3.2) | 24.9 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Participants recorded the occurrence of solicited local symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after product administration
Population: Population included all enrolled participants who received study product and provided safety data (via diary card and/or laboratory results) following vaccine administration (N=61). Two participants in Group 4B did not receive study product: for 1 participant, difficulties were experienced with vein access for blood sample collection, and 1 participant had a syncopal event during a blood draw.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  Pain/Tenderness: None | 4 | 12 | 9 | 8 | 0
  Pain/Tenderness: Mild | 1 | 3 | 6 | 5 | 11
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 2
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Swelling: None | 5 | 15 | 15 | 13 | 11
  Swelling: Mild | 0 | 0 | 0 | 0 | 2
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0
  Redness: None | 5 | 15 | 15 | 13 | 12
  Redness: Mild | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 1
  Pruritis (Itching): None | 5 | 15 | 15 | 13 | 12
  Pruritis (Itching): Mild | 0 | 0 | 0 | 0 | 1
  Pruritis (Itching): Moderate | 0 | 0 | 0 | 0 | 0
  Pruritis (Itching): Severe | 0 | 0 | 0 | 0 | 0
  Bruising: None | 5 | 15 | 15 | 13 | 13
  Bruising: Mild | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 4 | 12 | 9 | 8 | 0
  Any Local Symptom: Mild | 1 | 3 | 6 | 5 | 10
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 2
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Participants recorded the occurrence of solicited systemic symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  Malaise: None | 4 | 13 | 11 | 9 | 2
  Malaise: Mild | 1 | 2 | 4 | 4 | 8
  Malaise: Moderate | 0 | 0 | 0 | 0 | 3
  Malaise: Severe | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 5 | 14 | 14 | 12 | 4
  Myalgia: Mild | 0 | 1 | 1 | 1 | 7
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 2
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0
  Headache: None | 5 | 13 | 12 | 10 | 5
  Headache: Mild | 0 | 2 | 3 | 3 | 7
  Headache: Moderate | 0 | 0 | 0 | 0 | 1
  Headache: Severe | 0 | 0 | 0 | 0 | 0
  Chills: None | 4 | 14 | 15 | 12 | 3
  Chills: Mild | 1 | 1 | 0 | 1 | 8
  Chills: Moderate | 0 | 0 | 0 | 0 | 2
  Chills: Severe | 0 | 0 | 0 | 0 | 0
  Nausea: None | 5 | 14 | 14 | 13 | 10
  Nausea: Mild | 0 | 1 | 1 | 0 | 3
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): None | 5 | 15 | 15 | 13 | 10
  Temperature (Fever): Mild | 0 | 0 | 0 | 0 | 1
  Temperature (Fever): Moderate | 0 | 0 | 0 | 0 | 2
  Temperature (Fever): Severe | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 5 | 14 | 14 | 13 | 9
  Joint Pain: Mild | 0 | 1 | 1 | 0 | 4
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 4 | 12 | 10 | 7 | 1
  Any Systemic Symptom: Mild | 1 | 3 | 5 | 6 | 7
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0 | 5
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following Product Administration
Description: SAEs were recorded from receipt of product administration through the last study visit at Week 40. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after product administration through Day 280, up to Week 40
Population: Population included all enrolled participants who received study product (N=61). Two participants in Group 4B did not receive study product: for 1 participant, difficulties were experienced with vein access for blood sample collection, and 1 participant had a syncopal event during a blood draw.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 1 | 0 | 0 | 0
  Total Number of Participants who had SAE | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Product Administration
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of study product administration through the visit scheduled for 4 weeks after study product administration. At other time periods greater than 4 weeks after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module), influenza-like illness (ILI) or influenza and new chronic medical conditions that required ongoing medical management (reported as separate outcomes) were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 28 days post product administration, up to Week 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  Related to Study Product | 2 | 2 | 1 | 1 | 0
  Unrelated to Study Product | 2 | 6 | 5 | 2 | 7
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 4 | 8 | 6 | 3 | 7

5. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of study product administration through the last expected study visit at Week 40. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after product administration through Day 280, up to Week 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0 | 1
  Number of Participants With New Chronic Medical Condition | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following Product Administration
Description: Abnormal lab results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil percents/counts) and chemistry (alanine aminotransferase (ALT), alanine aspartate (AST), alkaline phosphate (ALP), creatinine and total bilirubin). Complete Blood Count (CBC) with differential, total bilirubin, AST, ALT, and ALP results were collected at Baseline, Day 0, Day 14, and 28. Creatinine results were collected at Baseline, Day 0 and Day 14. Institutional lab normal ranges as well as Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 through 28 days post product administration, up to Week 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  WBC Count | 1 | 0 | 0 | 0 | 0
  Bilirubin | 1 | 2 | 1 | 0 | 0
  Hemoglobin | 2 | 3 | 2 | 0 | 2
  Neutrophil Count | 2 | 0 | 0 | 0 | 0
  Lymphocyte Count | 0 | 0 | 0 | 1 | 1
  ALT | 0 | 1 | 0 | 0 | 0
  AST | 0 | 1 | 0 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 2 | 0 | 1 | 1 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 2 | 4 | 2 | 0 | 3
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 4 | 4 | 3 | 1 | 3

7. Primary Outcome: Number of Participants With Influenza or Influenza-like Illness (ILIs) Following Product Administration
Description: Influenza or influenza-like illness (ILI) were recorded in the study database from receipt of the study product administration through the last study visit. ILI was defined as fever (temperature of 100 degrees F [37.8 degrees C] or greater) and a cough and/or sore throat in the absence of a known cause other than influenza. Collection of nasopharyngeal swabs were used for laboratory confirmation of influenza by polymerase chain reaction (PCR) in participants who met criteria for ILI. Subsequently, results of any reported laboratory testing for identification of pathogens were included for cases meeting initial criteria for ILI. The severity of illness in participants with laboratory confirmed influenza illness were captured on a case report form rather than on an Adverse Event (AE) form.
Time Frame: Day 0 after product administration through Day 280, up to Week 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
Participants
  Reported Influenza-like Illness | 0 | 0 | 0 | 0 | 1
  Influenza confirmed by clinical test | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Antibody Response Following the Completion of Vaccination
Description: FluMos-v1-specific antibody titers were measured by Electrochemiluminescence Immunoassay (ECLIA) using a Meso Scale Discovery (MSD) platform. FluMos-v1 was biotinylated at an AviTag site located proximal to the C-terminus from the trimer foldon and bound to MSD streptavidin-coated plates. Serum samples collected at 2 weeks after product administration were assayed alongside healthy pooled human sera (not from this trial) as a reference standard. Binding of the reference standard to FluMos-v1 was assigned a stock concentration of 54000 arbitrary units per milliliter (AU/mL). Serial dilutions of sample within the dynamic range of the standard curve were interpolated to assign a sample concentration in AU/mL. Group geometric mean AU/mL values and 95% confidence intervals are reported.
Time Frame: Baseline to 2 weeks after product administration
Population: Population included all enrolled participants who received study product (N=61). Two participants in Group 4B did not receive study product: for 1 participant, difficulties were experienced with vein access for blood sample collection, and 1 participant had a syncopal event during a blood draw. Twelve (12) out of 13 participants were analyzed in Group 4 at Week 2 post administration, as serum was not collected for one Group 4 participant at Week 2.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
Number analyzed (Participants) | 5 | 15 | 15 | 13 | 13
AU/mL
  Week 0 Baseline (pre-administration) | 53182 [29435 to 96087] | 87179 [64657 to 117547] | 76775 [59572 to 98945] | 89289 [67820 to 117554] | 90907 [65566 to 126043]
  Week 2 (14 days after product administration): number analyzed (Participants) | 5 | 15 | 15 | 12 | 13
  Week 2 (14 days after product administration) | 76333 [43939 to 132610] | 160234 [117213 to 219045] | 114327 [91111 to 143458] | 142738 [115468 to 176450] | 241119 [188247 to 308841]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after product administration. Unsolicited AEs were recorded from receipt of product administration through the visit scheduled 4 weeks after administration. At other time periods greater than 4 weeks after administration, only serious AEs, influenza or influenza-like illness (ILI) and new chronic medical conditions that required ongoing medical management were recorded through study completion at Day 280.
Description: The overall Arms/Groups summarize AEs collected after product administration separately and grouped by the study product and dose. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity. Influenza/ILI were collected separately and not included as AE.
Arm/Group | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15 | 0/15 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/15 | 0/15 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/5 | 8/15 | 6/15 | 5/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) (N=5) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) (N=15) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) (N=15) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) (N=13) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v) (N=13)
Malignant oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Group 1 (1A-1B): FluMos-v1 (20 mcg) (N=5) | Part A, Group 2 (2A-2B): FluMos-v1 (60 mcg) (N=15) | Part A, Group 3 (3A-3B): Flucelvax (60 mcg) (N=15) | Part B, Group 4 (4A-4B): FluMos-v1 (100 mcg) (N=13) | Part B, Group 5 (5A-5B): FluMos-v1 (100 mcg) + Adjuplex (20% v/v) (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hangover (General disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Administration site pain (General disorders) | 1 | 3 | 6 | 5 | 13
Administration site swelling (General disorders) | 0 | 0 | 0 | 0 | 2
Chills (General disorders) | 1 | 1 | 0 | 1 | 10
Malaise (General disorders) | 1 | 2 | 4 | 4 | 11
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 4 — Joint Pain
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 7
Headache (Nervous system disorders) | 0 | 2 | 3 | 3 | 8
Administration site erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Administration site pruritis (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04896086/Prot_SAP_ICF_002.pdf